CLINICAL TRIAL: NCT00193908
Title: A Paired Double Blind Randomised Comparison of Cavilon(TM) Durable Barrier Cream(TM)[CDBC] to 10% Glycerine ("Sorbolene") Cream in the Prophylactic Management of Post-Mastectomy Irradiation Skin Care
Brief Title: Cavilon Breast Trial: Comparison of Cavilon Durable Barrier Cream to Glycerine ("Sorbolene") Cream
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: 3M (Industry)
Responsible Party: Dr Peter Graham, Trans Tasman Radiation Oncology Group (TROG)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TROG 04.01
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Breast Cancer
Keywords: Skin care; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cavilon (TM) Durable Barrier Cream; Drug: Sorbolene; Radiation: Radiotherapy
- 2 (Experimental)
  Interventions: Drug: Cavilon (TM) Durable Barrier Cream; Drug: Sorbolene; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cavilon (TM) Durable Barrier Cream — Cavilon (TM) Durable Barrier Cream will be applied to either the medial or the lateral side of the treated breast. Side will depend on randomisation.
Drug: Sorbolene — Sorbolene will be applied to either the medial or the lateral side of the treated breast. Side will be determined by randomisation
Radiation: Radiotherapy — Minimum prescribed dose to the chest wall is 45Gy in 25 fractions. Planning and Treatment is per the study protocol
  Other Names: Radiotherapy, Radiation Therapy

SUMMARY:
This study has patients using two different moisturising creams during radiation therapy after mastectomy. These are Cavilon and sorbolene. It is hypothesised that skin reactions may be reduced by the Cavilon cream compared to sorbolene.

DETAILED DESCRIPTION:
Skin reactions are a common and undesirable result of radiation treatment. Preventative measures are often used although there are few controlled trials. Commonly employed agents for established reactions have included sorbolene (10% Glycerine), silver sulphadiazine, hydrocolloid dressings, topical steroids, salt water or bicarbonate of soda water solution bathing and hydrogen peroxide. One trial found that Cavilon No-Sting Barrier film reduced Grade 3 skin reaction compared to sorbolene, although this film did not contain any moisturising agents.

General Hypothesis: That in a paired double blind randomised study peak and overall skin reactions experienced by post mastectomy breast cancer patients receiving radiotherapy may be reduced by Cavilon Durable Barrier Cream (CDBC) compared to Sorbolene.

Alternative Hypothesis of primary outcome: the frequency of grade 3 or more skin reaction will be reduced from 35% to 25% for skin care using sorbolene or CDBC respectively.

Alternative Hypothesis of secondary outcome: the mean area under the curve (AUC) of total skin reaction will be reduced from 9 to 8 for skin care using sorbolene or CDBC respectively.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or more years
* Post total mastectomy
* Planned dose at least 45 Gy in 25 fractions
* ECOG 0-2
* Able to attend weekly during treatment for review and photo and for up to 6 weeks after radiotherapy
* Patients capable of childbearing using adequate contraception
* Written informed consent

Exclusion Criteria:

* Previous radiotherapy to the chest wall to be treated
* Macroscopic cutaneous involvement by malignancy at time of radiotherapy
* Known allergy to product contents
* Patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2004-03; Primary Completion 2007-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Frequency of moist desquamation (grade 3) acute skin reaction scored as worst reaction within allocated skin care area | 12 weeks

SECONDARY OUTCOMES:
Skin toxicity area under the curve (AUC) being sum of maximum skin reaction per week over 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Graham, Study Chair — St George Hospital
Locations (12):
- Australia (12):
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Brisbane Hospital, Herston, Queensland
  - Mater QRI, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - Royal Perth Hospital, Perth, Western Australia

REFERENCES:
- [Derived] Graham PH, Plant N, Graham JL, Browne L, Borg M, Capp A, Delaney GP, Harvey J, Kenny L, Francis M, Zissiadis Y. A paired, double-blind, randomized comparison of a moisturizing durable barrier cream to 10% glycerine cream in the prophylactic management of postmastectomy irradiation skin care: trans Tasman Radiation Oncology Group (TROG) 04.01. Int J Radiat Oncol Biol Phys. 2013 May 1;86(1):45-50. doi: 10.1016/j.ijrobp.2012.12.009. Epub 2013 Feb 12. PMID 23414763
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au